CLINICAL TRIAL: NCT03315923
Title: Comparison of Expanded Disability Status Scale, Gad-enhanced Brain Lesions, Annualized Relapse Rate, and Side Effects Between Active Secondary Progressive Multiple Sclerosis Patients on Rituximab and Glatiramer Acetate
Brief Title: Comparison of Clinical Effects of Rituximab and Glatiramer Acetate in Secondary Progressive Multiple Sclerosis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vahid Shaygannejad, Professor of Neurology, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 396514
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Active secondary progressive Multiple Sclerosis; Glatiramer acetate; Rituximab; Comparative study; Disability; Randomized clinical trial; Annualized relapse rate
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Rituximab; Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental): Patients in this group will receive 1g of rituximab in 500 cc normal saline serum through intravenous infusion as one treatment course. The treatment course will be repeated in 6 months. Along with rituximab, 100 mg methylprednisolone, 10 mg chlorpheniramine, and 500 mg acetaminophen will also be injected to decrease side effects of rituximab.
  Interventions: Drug: Rituximab
- Glatiramer acetate (Experimental): Patients in this group will receive 40 mg of glatiramer acetate three times per week through subcutaneous injection.
  Interventions: Drug: Glatiramer Acetate

INTERVENTIONS:
Drug: Rituximab — Patients will receive 1 g of rituximab (two vials of Zytux 500 mg/50 ml) in 500 cc normal saline serum through intravenous infusion as one treatment cycle. This cycle will be repeated every 6 months. Along with rituximab, patients will receive 100 mg of methylprednisolone, 10 mg of chlorpheniramine, and 500 mg of acetaminophen. Before each cycle, patients will be evaluated regarding complete blood count (CBC)-diff, blood urea nitrogen (BUN), Cr, and liver function tests.
  Other Names: Zytux®
  Arms: Rituximab
Drug: Glatiramer Acetate — Patients will receive 40 mg of glatiramer acetate three times per week through subcutaneous injection. Patients will undergo electrocardiography before starting the treatment to find any abnormal finding. Also, lab tests will be checked for them prior to the treatment, including CBC-diff, BUN, Cr, and liver function tests.
  Other Names: Osvimer®
  Arms: Glatiramer acetate

SUMMARY:
The purpose of this study is to compare expanded disability status scale, annualized relapse rate, Gad-enhanced brain lesions, and side effects after administration of rituximab and glatiramer acetate among patients with active secondary progressive multiple sclerosis during a one year follow up through a randomized clinical trial.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune inflammatory demyelinative disease of central nervous system. Active secondary progressive MS means progressive accumulation of disability after an initial relapsing course which is also associated with clinical relapses and/or new/enlarged Gad-enhanced brain lesions. This form of the disease leads to high rates of morbidity and mortality among patients. Different immunosuppressive and immunomodulatory agents are recommended by researchers to decrease relapses and improve disability among MS patients. The effect of these medications on different phenotypes of MS are mostly investigated solely and very small number of comparative studies are conducted to evaluate the superiority of these medications on each other.

Glatiramer acetate is one of the known MS medications which is being used to control relapses from a long time ago and different clinical trials have shown its partial efficacy among MS patients. On the other hand, rituximab is one of the medications which is recently suggested for treatment of MS and currently phase II clinical trials are conducted to evaluate the efficacy of this medication among patients. As previously stated, there is a lack of clinical trials to compare the efficacy of suggested medications among secondary progressive patients. To fill this gap, we aimed to compare the efficacy of these two medications on disability, annualized relapse rate, and Gad-enhanced brain lesions among patients with active secondary progressive MS through a randomized clinical trial during a one-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years old
* diagnosis of active secondary progressive multiple sclerosis based on the latest McDonald criteria in 2010
* experiencing at least one relapse during the last year
* expanded disability status scale ≤5
* diagnosis of secondary progressive MS for at least one year
* maintaining pregnancy prevention methods for women in reproductive ages
* filling the written informed consent prior to enrollment

Exclusion Criteria:

* diagnosis of other subtypes of MS, including relapsing-remitting MS and primary progressive MS and inactive form of the disease
* experiencing relapse during the 30 days before starting the study
* receiving systemic corticosteroid therapy during the last 30 days
* undergoing plasmapheresis or receiving intravenous immunoglobulin during the last 1 months
* history of other demyelinative diseases of central nervous system such as neuromyelitis optica spectrum disorders
* history of other autoimmune diseases such as systemic lupus erythematosus, sjogren's syndrome, antiphospholipid syndrome, and behcet's disease
* presence of chronic or recurrent infections such as hepatitis B, hepatitis C, or syphilis
* pregnancy or lactation
* receiving live attenuated viral vaccines during the last 4 weeks
* history of cardiac arrhythmia, angina pectoris, or other cardiac diseases
* history of immunodeficiency syndromes such as HIV
* white blood cell count <2500 or lymphocyte count <400
* history of brain and spinal malignancies
* history of severe allergic reactions or anaphylaxis to monoclonal antibodies
* presence of active bacterial, viral, fungal, mycobacterial, or other infections
* alcohol or drug abuse during the last two years
* unable to undergo MRI
* presence of uncontrolled cardiac, respiratory, renal, hepatic, endocrine, or gastrointestinal disease
* presence of encephalopathy due to infectious (such as herpes, syphilis, ...) or metabolic (vitamin B12 deficiency) reasons
* history of bone marrow transplant, whole body radiotherapy, or other treatments leading to reduction of lymphocytes
* Cr>1.4 in women and >1.6 in men
* aspartate transaminase and alanine transaminase 2.5 times higher than the normal amount
* platelet count <100000
* Hb <8.5

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Disability measured by Expanded Disability Status Scale | one year
  expanded disability status scale will be measured in the baseline and after 12 months of intervention. This scale measures the disability of patients with a score, ranging from 0 (normal neurological exam) to 10 (death due to MS). This score is assigned to the patient by the neurologist and after neurological examination. The patient will be given a score in this scale according to the observed disability. The scores will be compared at the end of study.

SECONDARY OUTCOMES:
Adverse Drug Reactions | one year
  adverse drug reactions will be observed closely and reported during the intervention. We will compare the number of adverse drug reactions in two groups. Also, adverse drug reactions will be described by details in each group.
number of Gadolinium-enhanced brain lesions and neuroimaging findings | one year
  patients will undergo brain MRI before and after the study and number of Gad-enhanced brain lesions will compared before and after intervention.
Annualized relapse rate | one year
  annualized relapse rate will be measured in the baseline (according to patients' history in the last year) and after 12 months of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Vahid Shaygannejad, M.D., Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Kashani Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No
We may share the individual participant data (anonymously) on request of qualified investigators.

REFERENCES:
- [Background] Calabresi PA. Diagnosis and management of multiple sclerosis. Am Fam Physician. 2004 Nov 15;70(10):1935-44. PMID 15571060
- [Background] Leray E, Moreau T, Fromont A, Edan G. Epidemiology of multiple sclerosis. Rev Neurol (Paris). 2016 Jan;172(1):3-13. doi: 10.1016/j.neurol.2015.10.006. Epub 2015 Dec 21. PMID 26718593
- [Background] Hurwitz BJ. The diagnosis of multiple sclerosis and the clinical subtypes. Ann Indian Acad Neurol. 2009 Oct;12(4):226-30. doi: 10.4103/0972-2327.58276. PMID 20182569
- [Background] Tsang BK, Macdonell R. Multiple sclerosis- diagnosis, management and prognosis. Aust Fam Physician. 2011 Dec;40(12):948-55. PMID 22146321
- [Background] Wingerchuk DM, Carter JL. Multiple sclerosis: current and emerging disease-modifying therapies and treatment strategies. Mayo Clin Proc. 2014 Feb;89(2):225-40. doi: 10.1016/j.mayocp.2013.11.002. PMID 24485135
- [Background] Dhib-Jalbut S. Glatiramer acetate (Copaxone) therapy for multiple sclerosis. Pharmacol Ther. 2003 May;98(2):245-55. doi: 10.1016/s0163-7258(03)00036-6. PMID 12725872
- [Background] Schrempf W, Ziemssen T. Glatiramer acetate: mechanisms of action in multiple sclerosis. Autoimmun Rev. 2007 Aug;6(7):469-75. doi: 10.1016/j.autrev.2007.02.003. Epub 2007 Mar 6. PMID 17643935
- [Background] Khan O, Rieckmann P, Boyko A, Selmaj K, Ashtamker N, Davis MD, Kolodny S, Zivadinov R. Efficacy and safety of a three-times-weekly dosing regimen of glatiramer acetate in relapsing-remitting multiple sclerosis patients: 3-year results of the Glatiramer Acetate Low-Frequency Administration open-label extension study. Mult Scler. 2017 May;23(6):818-829. doi: 10.1177/1352458516664033. Epub 2016 Aug 8. PMID 27503905
- [Background] Mao CP, Brovarney MR, Dabbagh K, Birnbock HF, Richter WF, Del Nagro CJ. Subcutaneous versus intravenous administration of rituximab: pharmacokinetics, CD20 target coverage and B-cell depletion in cynomolgus monkeys. PLoS One. 2013 Nov 12;8(11):e80533. doi: 10.1371/journal.pone.0080533. eCollection 2013. PMID 24265828
- [Background] Bar-Or A, Calabresi PA, Arnold D, Markowitz C, Shafer S, Kasper LH, Waubant E, Gazda S, Fox RJ, Panzara M, Sarkar N, Agarwal S, Smith CH. Rituximab in relapsing-remitting multiple sclerosis: a 72-week, open-label, phase I trial. Ann Neurol. 2008 Mar;63(3):395-400. doi: 10.1002/ana.21363. PMID 18383069
- [Background] Hawker K, O'Connor P, Freedman MS, Calabresi PA, Antel J, Simon J, Hauser S, Waubant E, Vollmer T, Panitch H, Zhang J, Chin P, Smith CH; OLYMPUS trial group. Rituximab in patients with primary progressive multiple sclerosis: results of a randomized double-blind placebo-controlled multicenter trial. Ann Neurol. 2009 Oct;66(4):460-71. doi: 10.1002/ana.21867. PMID 19847908